CLINICAL TRIAL: NCT07244549
Title: Chronic Neurophyhsiological and Kinematic Biomarker Monitoring in Patients With Dystonia and Pallidal Deep Brain Stimulation
Brief Title: Chronic Outcome Monitoring for DBS in Dystonia
Acronym: COMMED
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other); Hannover Medical School (Other); Dystonia Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Dr Lucia K Feldmann, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: CCM_MDNS_COMMED-01
Record Dates: First submitted 2025-09-22; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Dystonia
Keywords: electrophysiology; biomarkers; deep brain stimulation; dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dystonia is a severe movement disorder involving increased muscular activity and can be very variable. To date, the treatment of dystonia is challenging. One effective therapy is deep brain stimulation (DBS), an invasive therapy, where stimulation electrodes are inserted in deep brain regions and a continuous electrical therapy is delivered via a pacemaker. However, the optimization of the therapy is a long process, up to months and there is no immediate adaptation to different disease states.

This project aims to improve DBS therapy: The first aim is to learn more about electrical brain activity that could be the feedback signal for individualized therapy. Secondly, the investigators want to gather information about the long-term development of the signal and potential hints for optimal therapy locations that could be acutely used to accelerate therapy optimization. To date, recordings mainly in lab settings, have suggested low-frequency activity as a biomarker for dystonia. Biomarkers are signals that are changed with therapy and that reflect symptom severity. Further understanding of the low-frequency biomarker for dystonia and its applicability in everyday life is one of the objectives in this study. Therefore, using a pacemaker that can also record brain activity, biomarker activity will be recorded for 12 months. At the same time, development of clinical symptoms will be assessed using an application with weekly questionnaires on symptoms and a video diary. At monthly appointments for data saving, resting state as well as motor activity during a finger tapping task will be recorded to also assess the development of side-effects, such as stimulation-induced slowing, and their biomarkers.

DETAILED DESCRIPTION:
Dystonia is a hyperkinetic movement disorder that can have various clinical phenotypes, from isolated cervical dystonia to severe generalized dystonia. Deep brain stimulation (DBS) is an effective therapy for dystonic symptoms and has been successfully used for more than 20 years. However, clinical optimization can be a complicated and lengthy process, and to date there is no closed-loop stimulation paradigm automatically adapting to current disease states.

Previous electrophysiological research using intracranial local field potential (LFP) recordings from DBS electrodes in the internal pallidal globe (GPi) has identified low-frequency activity in the theta/alpha band (7-12 Hz) as a physiomarker for symptom severity, although stimulation effects on the neurophysiology have only been investigated indirectly to date. Interestingly, stimulation-induced bradykinesia was correlated with increased beta-band activity, pointing towards transdiagnostic biomarkers. With the Percept neurostimulator (Medtronic Inc., Minnesota, USA) high resolution electrophysiological recordings, also during stimulation, and chronic biomarker tracking have become more accessible, also allowing for investigation of long-term dynamics such as circadian variations. To date, in dystonia, only case-reports have been published using this device.

Here, the development of electrophysiological biomarkers are systematically investigated during the first post-operative year. The aim is to, firstly, characterize the potential of low-frequency activity as a biomarker for adaptive algorithms. Secondly, neurophysiological signatures (e.g. low-frequency, gamma band activity) that are predictive of symptom improvement will be characterized, which might lead to electrophysiology-guided acceleration of therapy optimization.

All patients with dystonia, regardless of the dystonia type, between the age of 5-80 years, receiving surgery for pallidal deep brain stimulation electrode implantation and the Percept device are screened to participate in the study. Participants, and if applicable the legal guardians, will provide informed consent according to the ethics approval (EA1/164/23 and EA2/163/25). The aim is to include 20-30 patients with various types of dystonia.

The first dataset will be continuously recorded biomarker activity in the low-frequency range and beta band, to also assess development of stimulation-induced beta increases. Recordings will be done using the Percept Chronic BrainSense feature that allows for continuous assessment of peak biomarker activity at an investigator-selected peak at a 5 Hz window and a temporal resolution of one mean value/10min. For symptomatic correlation, subjective (patient reported outcome (PRO) questionnaire) and objective (video-based kinematic analysis) will be collected. The PRO will cover motor symptoms as well as non-motor symptoms such as mood and pain.

The second data set will be high-resolution local-field potential recordings at monthly lab visits. Here, different therapy states (ON/OFF DBS) will be recorded during rest (comfortably seated with open eyes) and a movement task (finger tapping). Additionally, standardized clinical scales such as the Burke-Fahn-Marsden-Dystonia-Rating Scale (BFMDRS) and the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) will be assessed by clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent for the study, or in pediatric patients, legal guardian or parent willing to give informed consent
* Diagnosis of dystonia, which may be isolated or generalized
* Wish to receive surgical intervention with DBS to the internal pallidal globe (GPi)
* Decision to receive the sensing-enabled neurostimulator (Percept neurostimulator) PC/RC
* Age 5-80 years

Exclusion Criteria:

* Severe psychiatric disorders (BDI>20)
* Other severe medical conditions, that may interfere with the successful paritcipation in the study protocol
* No consent given

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with dystonia who receive pallidal deep brain stimulation with the Percept IPG in the study centers are offered to participate in the study. Since dystonia is a variable condition that might also affect young patients, also children and youths will, together with their parents/legal guardians, be informed about the study and consented as possible.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Amount of low-frequency band oscillatory suppression | monthly recordings for 12 months
  Local field potential recordings of pallidal neuronal activity will be recorded using the Percept neurostimulator. On the one hand, automatically preprocessed peak-biomarker activty in the low-frequency range (7.8-12 Hz) will be recorded continuously using the Chronic BrainSense function of the Percept neurostimulator for one year at a temporal resolution of 1 sample/10 min. Over time and with optimization of clinical DBS settings, low frequency dynamics will change in correlation with symptom improvement.
  On the other hand, at monthly recordings, local field potentials at a sampling frequency of 250 Hz will be recorded ON and OFF stimulation at various intensities up to the therapeutic stimulation intensity. After preprocessing and transformation to the time-frequency domain, low frequency activity will be compared between different therapy settings.
Proportion of pathological increase in beta band oscillatory activity | monthly recordings for 12 months
  Local field potential recordings of pallidal neuronal activity will be recorded using the Percept neurostimulator. On the one hand, automatically preprocessed peak-biomarker activity in the beta band (13-35 Hz) will be recorded continuously using the Chronic BrainSense function of the Percept neurostimulator for one year at a temporal resolution of 1 sample/10 min. Over time and with chronic DBS settings, beta band activity will increase in correlation with development of bradykinesia.
  On the other hand, at monthly recordings, local field potentials at a sampling frequency of 250 Hz will be recorded ON and OFF stimulation at various intensities up to the therapeutic stimulation intensity. After preprocessing and transformation to the time-frequency domain, beta band activity will be compared between different therapy settings.

SECONDARY OUTCOMES:
Proportion of dystonic symptom improvement in patient reported outcomes | weekly, through study completion, up to 12 months
  Weekly patient reported outcomes focused on motor symptoms (4 items: general movement, walking, use of hands, neck muscle tenseness) will provide insights into subjective evaluation of participants, on a 9-points likert scale. Lower scores imply improved symptoms.
Proportion of dystonic symptom improvement in kinematic video-based analysis | weekly, through study completion, for up to 12 months
  Based on weekly video recordings or at least monthly recordings at the lab visits, automated models will be used to assess symptom severity. With DBS optimization, an improvement of symptom severity is expected, that can be objectified in video kinematics as angle of deviation from midline, smaller angles imply reduced deviation and symptom improvement.
Proportion of dystonic symptom improvement based on validated scales - Burke Fahn Marsden Dystonia Rating Scale | monthly, through study completion, for up to 12 months
  At the monthly recordings, trained clinicians and movement disorder specialists will assess the Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS), lower scores indicate symptom improvement.
Proportion of dystonic symptom improvement based on validated scales - Toronto Western Spasmodic Torticollis Rating Scale | monthly, through study completion, for up to 12 months
  At the monthly recordings, trained clinicians and movement disorder specialists will assess Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) in patients with cervical dystonia, lower scores indicate symptom improvement.
Proportion of non-motor symptom improvement | weekly, through study completion, for up to 12 months
  Weekly patient reported outcome questionnaires focused on non-motor symptoms, specifically on the symptoms wellbeing, mood, pain, stress, sleep, will provide insights into subjective evaluation of non motor symptoms, rated on a 9-points likert scale. Higher scores imply improved symptoms.
Rate of bradykinesia with velocity decrease | weekly, through study completion, for up to 12 months
  At the monthly recordings, finger tapping will be objectively recorded using accelerometry. With chronic DBS, the velocity of the tapping (m/s^2) will decrease.
Rate of bradykinesia with decreased acceleration | monthly, through study completion, for up to 12 months
  At the monthly recordings, finger tapping will be objectively recorded using accelerometry. With chronic DBS, the acceleration (g) in the measured accelerometry data will decrease.

OTHER OUTCOMES:
Unified Parkinson's Disease Rating Scale | at beginning and completion of the study, up to 12 months
  At the first recording (post-operatively) and the last recording (12 months post-surgery) the Unified Parkinson's Disease Rating Scale-III (UPDRS-III) is assessed. We expect a stimulation-induced increase (deterioration) of the UPDRS-III.
Beck's Depression Inventory | at beginning and end of study, up to 12 months
  At the first recording (post-operatively) and the last recording (12 months post-surgery) the Beck's Depression Inventory-II (BDI-II) is assessed. We expect a stimulation-associated reduction (=improvement) of the BDI-II.
Apathy Scale | at beginning and end of study, up to 12 months
  At the first recording (post-operatively) and the last recording (12 months post-surgery) the Starkstein Apathy Scale is assessed. We expect a stimulation-induced improvement of the Starkstein Apathy Scale.
Obsessive-Compulsive Symptoms | at beginning and end of study, up to 12 months
  At the first recording (post-operatively) and the last recording (12 months post-surgery) the Obsessive Compulsive Inventory (OCI) is assessed. We expect a stimulation-induced improvement of the OCI.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea A Kuehn, MD, Study Director — Charite University, Berlin, Germany
Locations (3):
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Heinrich Heine University, Düsseldorf, Nordrhein-Westfahlen
  - Charité Universitätsmedizin Berlin, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared upon reasonable requests and after completion of data sharing contracts through the Charité GDPR-approved data management platform Virtual Research Environment.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The Study Protocol will be made available upon request for potential collaborators, starting 16.08.2024 and beyond the study duration, as part of study publications and through the results section of the study registration.
  Analytic code will be made available through GitHub repositories along with the result publication process.

REFERENCES:
- [Background] Feldmann LK, Lofredi R, Neumann WJ, Al-Fatly B, Roediger J, Bahners BH, Nikolov P, Denison T, Saryyeva A, Krauss JK, Faust K, Florin E, Schnitzler A, Schneider GH, Kuhn AA. Toward therapeutic electrophysiology: beta-band suppression as a biomarker in chronic local field potential recordings. NPJ Parkinsons Dis. 2022 Apr 19;8(1):44. doi: 10.1038/s41531-022-00301-2. PMID 35440571
- [Background] Krause P, Mahlknecht P, Skogseid IM, Steigerwald F, Deuschl G, Erasmi R, Schnitzler A, Warnecke T, Muller J, Poewe W, Schneider GH, Vesper J, Warneke N, Eisner W, Prokop T, Muller JU, Volkmann J, Kuhn AA; Deep-Brain Stimulation for Dystonia Study Group. Long-Term Outcomes on Pallidal Neurostimulation for Dystonia: A Controlled, Prospective 10-Year Follow-Up. Mov Disord. 2025 Jun;40(6):1098-1111. doi: 10.1002/mds.30130. Epub 2025 Feb 5. PMID 39907392
- [Background] Kupsch A, Benecke R, Muller J, Trottenberg T, Schneider GH, Poewe W, Eisner W, Wolters A, Muller JU, Deuschl G, Pinsker MO, Skogseid IM, Roeste GK, Vollmer-Haase J, Brentrup A, Krause M, Tronnier V, Schnitzler A, Voges J, Nikkhah G, Vesper J, Naumann M, Volkmann J; Deep-Brain Stimulation for Dystonia Study Group. Pallidal deep-brain stimulation in primary generalized or segmental dystonia. N Engl J Med. 2006 Nov 9;355(19):1978-90. doi: 10.1056/NEJMoa063618. PMID 17093249
- [Background] Ledingham D, Gibbs M, Mills R, Jenkins A, Nicholson C, Hussain MA, Baker M, Pavese N. Decoding Cervical Dystonia: Insights from Local Field Potentials in a Case Study Utilizing Open-Source Toolboxes. Mov Disord Clin Pract. 2025 Oct;12(10):1675-1678. doi: 10.1002/mdc3.70164. Epub 2025 Jun 5. No abstract available. PMID 40470846
- [Background] Neumann WJ, Horn A, Ewert S, Huebl J, Brucke C, Slentz C, Schneider GH, Kuhn AA. A localized pallidal physiomarker in cervical dystonia. Ann Neurol. 2017 Dec;82(6):912-924. doi: 10.1002/ana.25095. Epub 2017 Dec 5. PMID 29130551
- [Background] Peach R, Friedrich M, Fronemann L, Muthuraman M, Schreglmann SR, Zeller D, Schrader C, Krauss JK, Schnitzler A, Wittstock M, Helmers AK, Paschen S, Kuhn A, Skogseid IM, Eisner W, Mueller J, Matthies C, Reich M, Volkmann J, Ip CW. Head movement dynamics in dystonia: a multi-centre retrospective study using visual perceptive deep learning. NPJ Digit Med. 2024 Jun 18;7(1):160. doi: 10.1038/s41746-024-01140-6. PMID 38890413
- [Background] Scheller U, Lofredi R, van Wijk BCM, Saryyeva A, Krauss JK, Schneider GH, Kroneberg D, Krause P, Neumann WJ, Kuhn AA. Pallidal low-frequency activity in dystonia after cessation of long-term deep brain stimulation. Mov Disord. 2019 Nov;34(11):1734-1739. doi: 10.1002/mds.27838. Epub 2019 Sep 4. PMID 31483903
- [Background] van Rheede JJ, Feldmann LK, Busch JL, Fleming JE, Mathiopoulou V, Denison T, Sharott A, Kuhn AA. Diurnal modulation of subthalamic beta oscillatory power in Parkinson's disease patients during deep brain stimulation. NPJ Parkinsons Dis. 2022 Jul 8;8(1):88. doi: 10.1038/s41531-022-00350-7. PMID 35804160